CLINICAL TRIAL: NCT07038590
Title: Use of Immersive Virtual Reality and Therapeutic Exercise as Complementary Therapy in Mild to Moderate Parkinson's Disease (InViPark): Multicenter Randomized Clinical Trial
Brief Title: Use of Immersive Virtual Reality and Therapeutic Exercise as Complementary Therapy in Mild to Moderate Parkinson's Disease (InViPark)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vigo (Other)
Responsible Party: Principal Investigator, Pablo Campo-Prieto, PhD, University of Vigo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HEALTHYFIT-UVIGO 1/2024; IISGS (Other: University of Vigo)
Record Dates: First submitted 2024-12-16; First posted 2025-06-26 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-06

CONDITIONS: Parkinson Disease (PD)
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual treatment in patient association (Active Comparator): Patients participate in memory, relaxation, and occupational therapy workshops.
  Interventions: Other: usual treatment patient association
- Exergame and virtual reality program + usual treatment (Experimental): Weekly sessions (2) of exergame with virtual reality added to the usual treatment
  Interventions: Other: exergame program with virtual reality; Other: usual treatment patient association

INTERVENTIONS:
Other: exergame program with virtual reality — Participants who attend a patient association will add to their usual therapies or virtual exercise program to be developed 2 days a week for 3 months.
  Arms: Exergame and virtual reality program + usual treatment
Other: usual treatment patient association — Common therapies in patient associations: memory workshops, relaxation, and occupational therapy

SUMMARY:
This document is intended to provide participant with information about a research study in which the participant is invited to participate. This study was approved by the Research Ethics Committee of ______________________________. If the participant decide to participate, will receive personalized information from the investigator. Please read this document beforehand, and the investigator will ask you any questions you may have to understand the details. If the participant wish, the participant can take this document, review it with others, and take your time to decide whether or not to participate. Participation in this study is completely voluntary and free of charge. The participant can decide not to participate, participate, or change your mind by withdrawing your consent at any time during the project without giving any explanation. The investigators assure the participant that this decision will not affect any future participation with this research group. What is the purpose of the study? To analyze whether the use of a physical exercise program in immersive virtual environments (video games) has greater positive effects on Parkinson's symptoms than traditional rehabilitation programs. Why is the participant being offered to participate? The participant is invited to participate because the participant is a person diagnosed with Parkinson's and because, within the Open Science policies of the University of Vigo, the Galicia Sur Biomedical Foundation, and the Nóvoa Santos Foundation, where bringing research closer to the reality of patients is emphasized, the investigators have selected the specialized Parkinson's center of which the participant is a member to participate in this study.

What does the participation consist of? The participation consists of carrying out 2/3 sessions per week on alternate days of physical exercise, and depending on whether the participant belong to the control or experimental group, the participant will do it regularly or recreated with a video game. The duration of each session will be 15 minutes. Be part of one group or another will depend on chance (like throwing a coin in the air and it comes up Heads or Cross). The total duration of the intervention in both cases is 3 months. During the project, 2 evaluations will be carried out: Initial evaluation and final evaluation. In all of them they will be collected information in relation to their pharmacological treatment linked to the pathology, autonomy functional balance, gait and risk of falls, functional balance, symptoms and disease monitoring and quality of life. Furthermore, in the experimental group the usability and security of the tool will be evaluated immersive virtual reality used. All these assessments will be carried out in your proximity center on the agreed day and time to optimize said process and will have an approximate duration of 30 minutes.

What discomforts or inconveniences does the participation have? The participation requires travel to your reference center to carry out the study. This program, like any physical activity or exercise, may involve greater tiredness and/or musculo-articular discomfort due to the type of exercise to which you will be subjected.

No relevant adverse effects have been recorded in the use of immersive virtual environments (video games).

DETAILED DESCRIPTION:
This document is intended to provide participant with information about a research study in which the participant is invited to participate. This study was approved by the Research Ethics Committee of ______________________________. If the participant decide to participate, will receive personalized information from the investigator. Please read this document beforehand, and the investigator will ask you any questions you may have to understand the details. If the participant wish, the participant can take this document, review it with others, and take your time to decide whether or not to participate. Participation in this study is completely voluntary and free of charge. The participant can decide not to participate, participate, or change your mind by withdrawing your consent at any time during the project without giving any explanation. The investigators assure the participant that this decision will not affect any future participation with this research group. What is the purpose of the study? To analyze whether the use of a physical exercise program in immersive virtual environments (video games) has greater positive effects on Parkinson's symptoms than traditional rehabilitation programs. Why is the participant being offered to participate? The participant is invited to participate because the participant is a person diagnosed with Parkinson's and because, within the Open Science policies of the University of Vigo, the Galicia Sur Biomedical Foundation, and the Nóvoa Santos Foundation, where bringing research closer to the reality of patients is emphasized, the investigators have selected the specialized Parkinson's center of which the participant is a member to participate in this study. What does the participation consist of? The participation consists of carrying out 2/3 sessions per week on alternate days of physical exercise, and depending on whether the participant belong to the control or experimental group, the participant will do it regularly or recreated with a video game. The duration of each session will be 15 minutes. Be part of one group or another will depend on chance (like throwing a coin in the air and it comes up Heads or Cross). The total duration of the intervention in both cases is 3 months. During the project, 2 evaluations will be carried out: Initial evaluation and final evaluation. In all of them they will be collected information in relation to their pharmacological treatment linked to the pathology, autonomy functional balance, gait and risk of falls, functional balance, symptoms and disease monitoring and quality of life. Furthermore, in the experimental group the usability and security of the tool will be evaluated immersive virtual reality used. All these assessments will be carried out in your proximity center on the agreed day and time to optimize said process and will have an approximate duration of 30 minutes. What discomforts or inconveniences does the participation have? The participation requires travel to your reference center to carry out the study. This program, like any physical activity or exercise, may involve greater tiredness and/or musculo-articular discomfort due to the type of exercise to which you will be subjected. No relevant adverse effects have been recorded in the use of immersive virtual environments (video games).

ELIGIBILITY:
Inclusion Criteria:

1. Suffering from idiopathic PD confirmed by a neurologist.
2. Presenting a stage between 1 and 3 on the Hoehn and Yahr scale.
3. Being able to move around unaided.
4. Absence of dementia with a score on the Mini-Mental State Examination (MMSE) of 18 or higher.
5. Being between 30 and 70 years of age.

Exclusion Criteria:

1. Comorbidity that makes physical exercise inadvisable and that prevents all scheduled assessments from being performed.
2. Severe visual and/or hearing disturbances that impede the session.
3. Having a history of vertigo, seizures, or epileptic seizures.
4. Presence of motor fluctuations and/or dyskinesias, gait blockages, or a history of recent falls.
5. Be receiving stable dopaminergic treatment without changes in the previous 3 months and with a prior plan not to change it during the duration of the study.
6. Be receiving second-line therapy (deep brain stimulation or intraduodenal pump).
7. Be participating in another clinical trial.
8. Not attend at least 80% of the immersive virtual reality sessions.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-09-05 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Falls | From start to end of treatment at 12 weeks
  Risk of falling measured with the Tinneti Test

SECONDARY OUTCOMES:
Functional Capacity: balance, gait and risk of falls | From start to end of treatment at 12 weeks
  Measured with the Tinnetti Test
Functional Capacity: gait function | From start to end of treatment at 12 weeks
  Measured with the Timed up and Go test
Functional Capacity: gait function in dual task | From start to end of treatment at 12 weeks
  Measured with the Timed up and Go-cog test
Functional Capacity: lower limbs strength | From start to end of treatment at 12 weeks
  Measured with the Five times sit to stand test
Functional Capacity: upper limbs strength | From start to end of treatment at 12 weeks
  Measured with the handgrip strength
Self-perceived quality of life | From start to end of treatment at 12 weeks
  The Parkinson's Disease Questionnaire (PDQ-39) assesses how often people with Parkinson's experience difficulties across 8 dimensions of daily living including relationships, social situations and communication. Range from 0 to 100, with higher scores indicating a lower quality of life.
Mood | From start to end of treatment at 12 weeks
  The BDI-II (Beck Depression Inventory-II) scale is used to assess the severity of depression in adults and adolescents. Range from 0 to 63, with higher scores indicating worse results
Symptoms of the disease | From start to end of treatment at 12 weeks
  The UPDRS Part III, also known as the motor examination, is a component of the Unified Parkinson's Disease Rating Scale (UPDRS). It assesses motor symptoms of Parkinson's disease, range 0-132 with a higher score indicating more severe motor impairment.
Cognitive ability | From start to end of treatment at 12 weeks
  The Mini-Mental State Examination (MMSE) score ranges from 0 to 30, with a higher score indicating better cognitive function.
Intrinsic aspects of exposure to virtual reality: cyber sickness | From start to end of treatment at 12 weeks
  SSQ is used for measuring users' level of sickness symptoms and is highly appreciated in VR research. Each item is rated with the scale from none, slight, moderate to severe. Through some calculations, four representative scores can be found. Nausea-related subscore (N), Oculomotorrelated subscore (O), Disorientation-related subscore (D) are the scores for the symptoms for the specific aspects. Total Score (TS) is the score representing the overall severity of cybersickness experienced by the users of virtual reality systems (1-48) high scores worse results
Intrinsic aspects of exposure to virtual reality: post game experiences | From start to end of treatment at 12 weeks
  GEQ can be applied after playing the game, several times over a longer period - also to see the changes in the experience. It is applicable for lab and field evaluation studies.Post game module - conserns experiences once a player has stopped gaming.Captures the game experience based on a number of items (such as positive affect, competence, immersion, flow, challenge) (0-4) high scores better results

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vigo, Pontevedra, Spain

IPD SHARING:
Plan to Share IPD: No